CLINICAL TRIAL: NCT04372953
Title: Positive End-Expiratory Pressure (PEEP) Levels During Resuscitation of Preterm Infants at Birth (The POLAR Trial).
Acronym: POLAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: University of Pennsylvania (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: POLAR #60303
Record Dates: First submitted 2020-04-27; First posted 2020-05-04 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Lung Injury; Preterm Birth
Keywords: Resuscitation; Positive End-Expiratory Pressure (PEEP); Bronchopulmonary Dysplasia
MeSH Terms: conditions — Lung Injury; Premature Birth; Bronchopulmonary Dysplasia | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Intervention Model Description: Two parallel group, non-blinded, 1:1 randomised controlled, multi-national, multi-centre, trial comparing dynamic PEEP ( dynamic group) with standard PEEP strategy (static group).
Who Masked: Outcomes Assessor
Masking Description: The clinical team within the Delivery Room managing enrolled and randomised infants will not be masked/blinded to the intervention.
  Members of the Research Team at participating sites will also not be masked/blinded to the intervention.
  Research staff based at the central Trial Coordinating Centre (TCC), the Data Coordinating Centre (DCCe) and the Trial Statistician will be blinded to assigned treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Static PEEP Group (Active Comparator): Delivery of PEEP at 5-6 cmH2O via a T-piece resuscitator using an initial fraction of inspired oxygen (FiO2) of 0.30 via local standard interface (facemask, nasopharyngeal tube or nasal prong). FiO2 and other aspects of respiratory care are then titrated using a standardised resuscitation algorithm.
  Interventions: Procedure: Positive End-Expiratory Pressure (PEEP)
- Dynamic PEEP Group (Experimental): Dynamic delivery of PEEP at 8 cmH2O via a T-piece resuscitator using an initial fraction of inspired oxygen (FiO2) of 0.30 via local standard interface (facemask, nasopharyngeal tube or nasal prong). PEEP levels increased step-wise to 10 and/or 12 cmH2O if FiO2/respiratory care needs to be escalated as per a standardised resuscitation algorithm.
  If an infant shows evidence of respiratory improvement during resuscitative care, PEEP will be reduced in a stepwise method by 2 cmH2O each reduction, but to no lower than 8 cmH2O.
  Interventions: Procedure: Positive End-Expiratory Pressure (PEEP)

INTERVENTIONS:
Procedure: Positive End-Expiratory Pressure (PEEP) — PEEP is the delivery of any level of positive pressure to the lungs during expiration, by any method of assisted respiratory support. As the intervention in the Delivery Room PEEP will be administered via any of:
  1. Continuous Positive Applied Pressure (CPAP; non-invasive respiratory support) During CPAP, no other type of positive pressure is delivered as the infant supports tidal ventilation using her/his own spontaneous breathing effort.
  2. Positive Pressure Ventilation (PPV) During PPV, PEEP is delivered between periods of an applied inflating pressure (PIP) delivered at a clinician-determined rate. PPV can be delivered via a mask or other non-invasive interface (also termed non-invasive positive pressure ventilation; NIPPV), or via an endotracheal tube (often termed continuous mechanical ventilation; CMV).

SUMMARY:
Premature babies often need help immediately after birth to open their lungs to air, start breathing and keep their hearts beating. Opening their lungs can be difficult, and once open the under-developed lungs of premature babies will often collapse again between each breath. To prevent this nearly all premature babies receive some form of mechanical respiratory support to aid breathing. Common to all types of respiratory support is the delivery of a treatment called positive end-expiratory pressure, or PEEP. PEEP gives air, or a mixture of air and oxygen, to the lung between each breath to keep the lungs open and stop them collapsing.

Currently, clinicians do not have enough evidence on the right amount, or level, of PEEP to give at birth. As a result, doctors around the world give different amounts (or levels) of PEEP to premature babies at birth.

In this study, the Investigators will look at 2 different approaches to PEEP to help premature babies during their first breaths at birth. At the moment, the Investigators do not know if one is better than the other. One is to give the same PEEP level to the lungs. The others is to give a high PEEP level at birth when the lungs are hardest to open and then decrease the PEEP later once the lungs are opened and the baby is breathing.

Very premature babies have a risk of long-term lung disease (chronic lung disease). The more breathing support a premature baby needs, the more likely the risk of developing chronic lung disease. The Investigators want to find out whether one method of opening the baby's lungs at birth results in them needing less breathing support.

This research has been initiated by a group of doctors from Australia, the Netherlands and the USA, all who look after premature babies.

DETAILED DESCRIPTION:
All infants born <29 weeks' postmenstrual age (PMA) require positive end-expiratory pressure (PEEP) at birth. PEEP is a simple, feasible and cost-effective therapy to support extremely preterm infants that is used globally. The effective and safe level of PEEP to use after preterm birth remains the most important unanswered question in neonatal respiratory medicine.

The Investigators will undertake an international multi-centre randomised controlled trial to address in extremely preterm infants, whether the use of a high, dynamic PEEP level strategy to support the lung during stabilisation ('resuscitation') at birth, compared to the current practice of a static PEEP level, will reduce the rate of death or bronchopulmonary dysplasia (BPD).

This trial will address the following four key knowledge gaps:

1. Assessing whether individualising (dynamic) PEEP is superior to static PEEP
2. The uncertainty regarding applied pressure strategies to support the lung during stabilisation at birth arising from the lack of a properly powered, well-designed randomised trial specifically addressing important outcomes for respiratory support in the Delivery Room
3. The optimal PEEP strategy to use
4. Determining the differential effects of PEEP at different gestational ages.

For this study, the term PEEP refers to the delivery of positive pressure (via a bias flow of gas) to the lungs during expiration by any method of assisted respiratory support, this includes:

1. Continuous Positive Applied Pressure (CPAP; a method of non-invasive respiratory support). During CPAP no other type of positive pressure is delivered as the infant supports tidal ventilation using her/his own spontaneous breathing effort. PEEP during CPAP has also been called 'continuous distending pressure.
2. Positive Pressure Ventilation (PPV). During PPV PEEP is delivered between periods of an applied inflating pressure (PIP) delivered at a clinician-determined rate. PPV can be delivered via a mask or other non-invasive interface (also termed non-invasive positive pressure ventilation; NIPPV), or via an endotracheal tube (often termed continuous mechanical ventilation; CMV).
3. High-frequency oscillatory ventilation (HFOV) or high-frequency jet ventilation. These are modes of invasive PPV in which PIP is delivered at very fast rates (>120 inflations per minute) and at very small tidal volumes. During HFOV a mean airway pressure is determined by the clinician which is equivalent to the PEEP during other modes. During high-frequency jet ventilation the clinician sets a PEEP similar to CMV.

As all of these modes of ventilation have a similar goal of applying a pressure to the lung during expiration (usually to prevent lung collapse) the term PEEP has the same physiological result despite different methods of application.

The specific aim of the trial is to establish whether the use of a high, dynamic 8-12 cmH2O PEEP level ('dynamic') strategy to support the lung during stabilisation at birth, compared with a static 5-6 cmH2O PEEP level ('static') strategy, increases the rate of survival without bronchopulmonary dysplasia (BPD) in extremely preterm infants born <29 weeks' PMA, and reduces rates of common neonatal morbidities.

The Investigators hypothesise that in preterm infants born <29 weeks PMA who receive respiratory support during stabilisation at birth, a high, dynamic PEEP strategy (i.e. PEEP 8-12 cmH2O individualised to clinical need) as compared to a standard, static PEEP of 5-6 cmH2O, will:

1. Increase survival without BPD (primary outcome); and
2. Reduce rates of common neonatal morbidities such as failure of non-invasive respiratory support in the first 72 hours of life (secondary outcome).

This trial is a phase III/IV, two parallel group, non-blinded, 1:1 randomised controlled, multi-national, multi-centre study comparing dynamic PEEP (dynamic group) with standard PEEP strategy (static group).

The intervention will take place in the Delivery Room. The intervention period will be from the time of birth until 20 minutes of life or transfer from Delivery Room to NICU (whatever comes first). The follow-up period will extend to 36 weeks PMA (primary endpoint), and 24 months corrected GA to determine important long-term neurodevelopmental and respiratory outcomes.

The clinical team within the Delivery Room managing enrolled and randomised infants will not be masked/blinded to the intervention. Clinicians need to be able to see the PEEP delivery device to assess efficacy of pressure delivery. The Research Coordinator/Study team at site will also not be masked/blinded to the intervention, as they will be entering trial data into the data management system.

Research staff based at the central Trial Coordinating Centre (TCC), the Data Coordinating Centre (DCCe) and the trial statistician will be blinded to assigned treatment.

There will be a total of 906 infants recruited (453 in the Dynamic group, 453 in the Static group), over 25 recruitment centres across Australia, Europe, the United Kingdom, the Middle East, Canada and North America.

The study will have Regional Coordinating Centres (RCCs) established in the following jurisdictions:

1. Australia - The Murdoch Children's Research Institute/Royal Women's Hospital, Melbourne, AUS
2. The Netherlands - Amsterdam University Medical Centre, Netherlands, EU
3. The United Kingdom - The University of Oxford / National Perinatal Epidemiology Unit (NPEU), Oxford, UK, and
4. North America - the Hospital of the University of Pennsylvania, Pennsylvania, USA.

ELIGIBILITY:
Inclusion Criteria:

* Infants born between 23 weeks 0 days and 28 weeks 6 days PMA (by best obstetric estimate).
* Receives respiratory intervention (resuscitation) at birth with CPAP and/or positive pressure ventilation in the Delivery Room, to support transition and/or respiratory failure related to prematurity.
* Has a parent or other legally acceptable representative capable of understanding the informed consent document and providing consent on the participant's behalf either prospectively or after birth and randomisation if prenatal consent was not possible (at sites where the Ethics Committee permits waiver of prospective consent).

Exclusion Criteria:

* Not for active care based on assessment of the attending clinician or family decision
* Anticipated severe pulmonary hypoplasia due to rupture of membranes <22 weeks with anhydramnios or fetal hydrops
* Major congenital anomaly or anticipated alternative cause for respiratory failure
* Refusal of informed consent by their legally acceptable representative
* Does not have a guardian who can provide informed consent.

Ages: 23 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 906 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
The prevalence of the composite outcome of either death or bronchopulmonary dysplasia (BPD), as assessed by standard oxygen reduction test. | At 36 weeks post menstrual age.
  This is defined as the proportion of participants in the analysis set with a confirmed death date or a diagnosis of bronchopulmonary dysplasia (BPD), at 36 weeks post menstrual age.

SECONDARY OUTCOMES:
The rate/incidence of failure of non-invasive ventilation in first 72 hours, as assessed by intubation status. | From the time of birth until 72 hours post birth.
  This is defined as the proportion of participants in the analysis set requiring invasive ventilation (i.e. insertion of a Endotracheal Tube (ETT) within the first 72 hours after birth.
The rate/incidence of death within the first 10 days of life, as assessed by date of death. | From the time of birth until 10 days post birth.
  This is defined as the proportion of participants in the analysis set having dies within the first 10 days post birth.
Oxygen requirement ≥50% for 3 or more consecutive hours in first 72 hours | From the time of birth until 72 hours post birth.
  This is defined as highest FiO2 applied for 3 or more consecutive hours in the first 72 hours of age.
Supplementary oxygen use | From the time of birth until 10 days of age.
  This is defined as highest FiO2 in the delivery room, and then at 24 hours, 72 hours, 7 days and 10 days of age.
The rate/incidence of surfactant therapy requirement within the first 72 hours of life, as assessed by surfactant therapy status. | From the time of birth until 72 hours post birth.
  This is defined as the proportion of participants in the analysis set requiring surfactant therapy within the first 72 hours post birth.
The rate/incidence of grade 3 and 4 intraventricular haemorrhage within the first 72 hours of life, as defined via imaging. | From the time of birth until 72 hours post birth.
  This is defined as the proportion of participants in the analysis set requiring experiencing a grade 3 or 4 intraventricular haemorrhage, within the first 72 hours post birth.
The rate/incidence of treatment failure within the delivery room, as assessed by intubation status. | From the time of birth through transfer to NICU (within two hours from birth)
  This is defined as the proportion of participants in the analysis set requiring intubation (i.e. insertion of a Endotracheal Tube (ETT) within the delivery room, but prior to transfer to NICU.
The grade of bronchopulmonary dysplasia (BPD), based on the results of an oxygen reduction test. | At 36 weeks post menstrual age.
  This is defined as the grade bronchopulmonary dysplasia (BPD) assigned according to the results of an oxygen reduction test and mode or respiratory support at 36 weeks PMA (see Jensen et al Am J Resp Crit Care Med 2019;200:751-759).
Incidence of Death at 36 week PMA | At 36 weeks post menstrual age.
  This is defined as death at 36 weeks PMA (individual component of primary outcome)
Incidence of Bronchopulmonary dysplasia (BPD) at 36 week PMA | At 36 weeks post menstrual age.
  This is defined as the incidence of BPD at 36 weeks PMA (individual component of primary outcome)
Incidence of air leak and/or pulmonary interstitial emphysema (defined on chest radiograph; CXR) in the first 10 days after birth | Birth to 10 days of age.
  Any airleak, defined as Pneumothorax, pulmonary interstitial emphysema and/or pneumomediastimum, diagnosed by chest radiology within the first 10 days after birth.
Airleak | During hospital stay, on average until 36 weeks PMA.
  Any airleak, defined as Pneumothorax, pulmonary interstitial emphysema and/or pneumomediastimum, diagnosed by chest radiology. Airleak will be coded as occurring in the delivery room, in first 10 days of life, during hospital stay and if requiring drainage (e.g. via a chest tube)
Retinopathy of prematurity (stage 3 or higher or requiring treatment) | 36-week corrected PMA.
  Defined as retinopathy of prematurity (stage 3 or higher or requiring treatment) diagnosed by ophthalmological examination at or before 36-week corrected PMA
Significant brain injury (IVH grade 3 or 4, periventricular leukomalacia) | 36-week corrected PMA.
  Significant brain injury (IVH grade 3 or 4, periventricular leukomalacia) at or before 36-week corrected PMA as assessed by ultrasound or MRI cranial imaging.
Invasive ventilation at day 10 of age | First 10 days after birth.
  The rates of invasive ventilation (placement of an endotracheal tube for >4 hours) by day 7 and 10 of age
Highest PEEP used during non-invasive ventilation | Birth to 10 days of age.
  Defined as the highest PEEP used during non-invasive ventilation in the NICU (after delivery room management) at 24 hours, 72 hours, 7 and 10 days of age.
Duration of respiratory support | 36 week PMA.
  Defined as the total number of days of all forms of respiratory support (supplementary oxygen therapy, non-invasive and invasive ventilation)
Postnatal steroid use | 36 week PMA.
  Defined as the incidence of one or more course of postnatal steroids for the treatment of BPD
Inotrope use | 36 week PMA.
  Defined as the incidence of the administration of one or more inotropic agent by continuous infusion (not as a resuscitative agent) for more than 1 hour.
Length of stay in hospital | Up to 44 weeks PMA
  Defined as the total number of completed days in hospital related to the initial admission for management of preterm birth.
Oxygen requirement at discharge to home | Up to 44 weeks PMA
  Defined as the incidence of infants being discharged home on any form of oxygen therapy
Patent ductus arteriosus requiring medical or surgical therapy in first 72 hours | 72 hours of age.
  Defined as the incidence of patent ductus arteriosus requiring medical or surgical therapy in first 72 hours
Meeting the protocol criteria for failure of non-invasive ventilation during the intervention period | Up to the first 20 minutes after commencing respiratory support following birth.
  This is defined as the proportion of participants in the analysis set who met the criteria for requiring invasive ventilation (i.e. insertion of a Endotracheal Tube (ETT) within the first 72 hours after birth.

CONTACTS AND LOCATIONS:
Overall Officials: David Tingay, MBBS FRACP, Principal Investigator — Royal Children's Hospital
Locations (28):
- United States (4):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sharp Mary Birch Hospital for Women & Newborns, San Diego, California
  - Indiana University / Riley Children Health at Indiana University Health, Indianapolis, Indiana
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
- Australia (5):
  - Mater Misericordiae, South Brisbane, Queensland
  - Women & Childrens Hospital Adelaide, Adelaide, South Australia
  - Joan Kirner Women & Children's Hospital - VIC, Melbourne, Victoria
  - The Royal Women's Hospital, Melbourne Australia, Parkville, Victoria
  - King Edward Memorial Hospital, Subiaco, Western Australia
- Academic Teaching Hospital, Feldkirch, Feldkirch, Austria
- Antoine Beclere Medical Center / South Paris University Hospitals, Paris, Paris, France
- Italy (6):
  - Careggi Hospital, Florence, Florence
  - Ospedale Maggiore Policlinico, Milan, Milan
  - Vittore Buzzi Children's Hospital / Ospedale dei Bambini, Milan, Milan
  - San Gerardo Hospital, Monza, Milan
  - Filippo del Ponte Hospital, Varese, Milan
  - Gemelli University Hospital, Rome, Rome
- Netherlands (3):
  - Amsterdam University Medical Centre, Amsterdam, Amsterdam
  - Amalia Children's Hospital Radboudumc, Nijmegen, Nijmegen
  - Maxima Medical Centre, Veldhoven, Veldhoven
- Poznan University of Medical Sciences, Poznan, Poznan, Poland
- United Kingdom (7):
  - Birmingham Heartlands Hospital, Birmingham, England
  - Southmead Hospital, Bristol, England
  - James Cook University Hospital, Middlesbrough, England
  - Royal Infirmary Edinburgh, Edinburgh, Scotland
  - Royal Hospital for Children, Glasgow, Scotland
  - University Hospital Wishaw, Wishaw, Scotland
  - University Hospitals Leicester, Leicester

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for this analysis of the POLAR trial will be available six months after publication of the primary outcome.
  The study protocol, statistical analysis plan and consent forms will also be available. The data may be obtained from the Murdoch Children's Research Institute by emailing david.tingay@rch.org.au and mctc@mcri.edu.au.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication of primary outcome.
Access Criteria: Prior to releasing any data the following are required:
  1. A Data Transfer Agreement must be signed between relevant parties.
  2. The MCRI Sponsorship Committee must review and approve your protocol and statistical analysis plan which must include and describe how the data will be used and analysed.
  3. An Authorship Agreement to be agreed to and signed between relevant parties. The Agreement must include details regarding appropriate recognition. Authorship may not be justifiable but some form of acknowledgement is requested.
  4. Agreement to cover any additional costs relating to the provision of the data.
  5. Evidence of ethics approval or waiver of approval, to be compliant with the data transfer agreement and ethics requirements at our end.
  Data will only be shared with a recognised research institution where the MCRI Sponsorship Committee has approved the proposed analysis plan.
URL: https://www.melbournechildrens.com/mctc/

REFERENCES:
- [Background] Jensen EA, Dysart K, Gantz MG, McDonald S, Bamat NA, Keszler M, Kirpalani H, Laughon MM, Poindexter BB, Duncan AF, Yoder BA, Eichenwald EC, DeMauro SB. The Diagnosis of Bronchopulmonary Dysplasia in Very Preterm Infants. An Evidence-based Approach. Am J Respir Crit Care Med. 2019 Sep 15;200(6):751-759. doi: 10.1164/rccm.201812-2348OC. PMID 30995069